CLINICAL TRIAL: NCT00797654
Title: Integrated HIV Prevention and Trauma Treatment in MSM With Sexual Abuse History (Project THRIVE)
Brief Title: HIV Prevention and Trauma Treatment in Men Who Have Sex With Men and Who Have a History of Sexual Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenway Community Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Conall O'Cleirigh, Assistant Professor, Harvard Medical School, Director, Behavioral Medicine, Department of Psychiatry Massachusetts General Hospital, Fenway Community Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH081760-02 (NIH); R34MH081760-02 (NIH)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Risk Reduction
Keywords: Sexual Risks for HIV; Psychosocial Sequelae Relating to Childhood Sexual Abuse
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive pre and post HIV-test counseling and an information-motivation-behavior skills training combined with cognitive processing therapy
  Interventions: Behavioral: Information-motivation-behavior skills and cognitive processing therapy; Behavioral: Pre and Post HIV-Test Counseling
- 2 (Active Comparator): Participants will receive pre and post HIV-test counseling
  Interventions: Behavioral: Pre and Post HIV-Test Counseling

INTERVENTIONS:
Behavioral: Information-motivation-behavior skills and cognitive processing therapy — Treatment will include elements from effective interventions for reducing risky sexual behaviors and reducing post-traumatic stress disorder (PTSD) symptoms.
  Arms: 1
Behavioral: Pre and Post HIV-Test Counseling — Treatments are aimed at assessing and reducing behaviors that put participants at high risk of HIV infection.

SUMMARY:
This study will develop a therapy for men who have sex with men who also have a history of childhood sexual abuse to reduce behaviors that put them at a high risk of HIV infection.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) represent the largest group of new HIV infections. Rates of childhood sexual abuse (CSA) in MSM have been estimated to be higher than in the rest of the population, with some researchers estimating that 37% of all MSM have experienced CSA. CSA in MSM is associated with both higher rates of HIV risk behavior and higher rates of HIV infection. Treatments for preventing HIV are also less likely to be effective in MSM with a history of CSA, and these individuals tend to have higher rates of depression, anxiety, substance abuse, and post-traumatic stress disorder (PTSD) symptoms. This study will create and then test a new HIV prevention therapy that addresses both HIV risk behaviors and the co-occurring psychological health problems in MSM with a history of CSA.

This study includes a pilot phase and an experimental phase. In the pilot phase, the therapeutic treatment will be developed based on elements of successful interventions for reducing sexual risk-taking behaviors and PTSD symptoms. Information-motivation-behavioral (IMB) skills training for sexual risk reduction will be the basis for one of two treatment components, and it is expected to last for two 50-minute sessions. This intervention will include addressing knowledge about issues surrounding sexual risk, using motivational interviewing to address goals and self-efficacy, and providing strategies for behavioral change. Cognitive processing therapy (CPT) for CSA will be the basis for the other component and is expected to last for eight 50-minute sessions. Elements of this intervention will include identifying sexual abuse events, learning how to identify cognitive distortions, and learning processes to challenge and process these distortions.

During the pilot phase, approximately 10 participants will undergo the new treatment. After completing the treatment sessions, participants will undergo exit interviews, in which researchers will solicit feedback about the strengths and weaknesses of the treatment. This feedback will be used to fine tune the treatment.

During the second phase of the study, approximately 50 individuals will be randomly assigned to receive either HIV testing with pre/post-test counseling alone or in combination with the newly developed treatment. The experimental, integrated treatment will be administered over 10 individual therapy sessions comprised of sexual risk reduction counseling and cognitive therapy.

All participants will undergo assessments at enrollment and after treatment (or approximately 3 months after enrollment in comparator group), and at follow-up visits 6 and 9 months after enrollment. These assessments will measure sexual risk behaviors, PTSD symptoms, distress, social support, and substance abuse. Brief questionnaires about sexual behavior and measures of distress will be administered during the integrated treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as a biological man who has sex with men
* Reports history of childhood sexual abuse (sexual contact before the age of 13 with an adult or person 5 years older or sexual contact with the threat of force or harm between the ages of 13 and 16, inclusive, with a person 10 years older)
* Reports unprotected anal or vaginal intercourse within the past 3 months
* HIV-negative serostatus
* Able to understand English

Exclusion Criteria:

* All episodes of unprotected anal or vaginal intercourse occurred with only a single, primary HIV-negative partner
* Significant mental health diagnosis requiring immediate treatment, such as acute major depression, panic disorder, or any psychotic disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Self-reported sexual risk taking | Measured pre- and post-treatment and after 6 and 9 months
  For both the Treatment (Cognitive Processing Therapy with Information Motivation Behavior) and Control arms, participants will self-report sexual risk taking at baseline, 3-month post baseline, and at 6 and 9-month follow-ups (after enrollment).

SECONDARY OUTCOMES:
Reductions in negative effects of trauma, with cognitive and behavioral variables tested as potential mediators of treatment outcome | Measured pre- and post-treatment and after 6 and 9 months
  As with the baseline assessment, the Davidson Post-Traumatic Stress Disorder scale, and the MINI Neuro-psychiatric Interview for PTSD will be administered by an Independent Assessor who will be blind to participant group assignment.

CONTACTS AND LOCATIONS:
Overall Officials: Conall M. O'Cleirigh, PhD, Principal Investigator — Fenway Community Health
Locations (2):
- United States (2):
  - Fenway Community Health, Boston, Massachusetts
  - Fenway Health, Boston, Massachusetts